CLINICAL TRIAL: NCT01546155
Title: The Influence of Pressure Pain on [11C]Diprenorphine Binding Potentials
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jian Kong, Assistant Professor, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2011P0022171
Record Dates: First submitted 2012-02-24; First posted 2012-03-07 (Estimated); Results first posted 2017-04-11 (Actual); Last update posted 2017-04-11 (Actual); Status verified 2017-01

CONDITIONS: Healthy Controls
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- healthy controls (Experimental)
  Interventions: Radiation: PET imaging

INTERVENTIONS:
Radiation: PET imaging — Up to a 120 minute PET scan using [11C]diprenorphine as the radiotracer

SUMMARY:
Healthy volunteers aged 21 to 50 are needed for a research study investigating whether pain will alter the binding properties of ([11C]diprenorphine), a molecule that can be used during brain imaging. Positron Emission Tomography (PET) and functional Magnetic Resonance (fMRI) imaging will be used in this study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female adults, 21 to 50 years of age
* No contraindications to fMRI and PET scanning
* Within 15% of ideal body mass index (BMI)

Exclusion Criteria:

* Current significant medical, neurological, or psychiatric illness as assessed by the Physician Investigators
* Women who are pregnant or breast feeding, have gone through menopause, and/or have irregular menstrual cycles
* Claustrophobia
* History of head trauma
* Instability of responses to experimental pain (See Study Procedure Section Part II)
* History of asthma
* Use of psychotropic drugs or hormone treatments (including hormonal birth control) within one year of date of consent
* History of smoking
* Routine exercise in excess of one hour per day and/or three times per week
* Non-fluent English speaker

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2011-12; Primary Completion 2012-10 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jian Kong, MD (equiv), MS, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Charlestown, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Volunteers: The PET/fMRI scan session will last up to 120 minutes. Subjects will have 2 MR-PET scan sessions, each lasting up to 120 minutes, with a break between scan sessions. Approximately nine venous blood samples will be taken per scan session with a maximum of 48mL of blood drawn per scan session. Intermittent cuff pain, based on the previously determined Strong ratings, will be applied during one of the two scan sessions. Subjects will rate the pain they feel as a result of the cuff stimuli using the Gracely scale.
Period: Overall Study
Arm/Group | Healthy Volunteers
Started | 11
Completed | 8
Not Completed | 3
Not completed — could not tolerate long scan duration | 3

BASELINE CHARACTERISTICS:
Groups:
- Healthy Volunteers: The PET/fMRI scan session will last up to 120 minutes. Subjects will have 2 MR-PET scan sessions, each lasting up to 120 minutes, with a break between scan sessions. Approximately nine venous blood samples will be taken per scan session with a maximum of 48mL of blood drawn per scan session. Intermittent cuff pain, based on the previously determined Strong ratings, will be applied during one of the two scan sessions. Subjects will rate the pain they feel as a result of the cuff stimuli using the Gracely scale. The additional scan session for subjects will be performed under no pain, "control" conditions.
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.1 (2.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: PET/MRI Brain Activation
Description: Simultaneously collect fMRI-PET data in humans to investigate the change between bold signal evoked by pressure pain and bold signal evoked by non-painful pressure.
  The PET analyses generates one value per 120 minutes. This value is compared to the other 120 minute scan PET value in order to reflect the change.
Time Frame: day one
Measure: Mean (Standard Deviation); unit: percentage BOLD signal change
Arm/Group | Healthy Controls
Number analyzed (Participants) | 8
percentage BOLD signal change | 0.21 (0.13)

ADVERSE EVENTS:
Groups:
- Healthy Volunteers: PET imaging: Up to a 120 minute PET scan using [11C]diprenorphine as the radiotracer
Arm/Group | Healthy Volunteers
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No